CLINICAL TRIAL: NCT07206823
Title: An Open-label, Single-arm, Single-center Study to Evaluate the Efficacy and Safety of Romiplostim N01 in Combination With Rituximab in Patients With Primary Immune Thrombocytopenia Refractory to Oral TPO-RAs
Brief Title: Efficacy and Safety of Romiplostim N01 Combined With Rituximab in Patients With Oral TPO-RA-Refractory Primary Immune Thrombocytopenia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025767
Record Dates: First submitted 2025-09-26; First posted 2025-10-03 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-09

CONDITIONS: Primacy Immune Thrombocytopenia
MeSH Terms: interventions — Rituximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Romiplostim N01 + Rituximab Combination Therapy (Experimental)
  Interventions: Drug: Romiplostim N01; Drug: Rituximab

INTERVENTIONS:
Drug: Romiplostim N01 — Romiplostim N01 will be administered via subcutaneous injection once weekly based on the platele count. The starting dose is set at 3 μg/kg. Weekly dose adjustments will be guided by platelet counts measured immediately prior to administration, as follows:
  For a platelet count below 50 × 10⁹/L, the dose will be increased by 1 μg/kg.
  For a platelet count between 50 and 200 × 10⁹/L, the current dose will be maintained as the minimum therapeutic dose for bleeding risk reduction.
  For a platelet count between 200 and 400 × 10⁹/L, the dose will be decreased by 1 μg/kg.
  For a platelet count exceeding 400 × 10⁹/L, the administration will be withheld. It is stipulated that dosing will resume at a reduction of 1 μg/kg from the previous dose once the platelet count returns to 200 × 10⁹/L or below.
  Under no circumstances shall the dose exceed the maximum allowable limit of 10 μg/kg per week.
Drug: Rituximab — Rituximab will be administered in accordance with the Chinese guidelines for the diagnosis and management of adult primary immune thrombocytopenia (2020 edition). The dosage will be 375 mg/m² per infusion, administered via intravenous infusion once weekly for a total of four weeks.

SUMMARY:
The primary objective of this trial is to assess the efficacy and safety of combining Romiplostim N01 with Rituximab for the treatment of adult patients with primary immune thrombocytopenia (ITP) whose disease is refractory to oral TPO-RAs.

All participants in this study will receive the same combination treatment:

Rituximab: Given once a week through an intravenous infusion for 4 weeks. Romiplostim N01: Given as a weekly injection，the dose may be adjusted each week based on the patient's platelet count.

Participants will be asked to:

Visit the clinic regularly for check-ups, blood tests (to monitor platelet counts), and safety assessments.

Report their bleeding symptoms for evaluation. This is an open-label, single-arm trial, meaning that all participants will receive the investigational treatment, and both the research team and participants will be aware of the treatment assigned. The study aims to enroll approximately 30 adult patients aged 14 years or older who have been diagnosed with ITP and have not responded adequately to prior oral TPO-RAs (eltrombopag/hetrombopag).

ELIGIBILITY:
Inclusion Criteria:

Confirmed diagnosis of primary immune thrombocytopenia (ITP).

Age ≥14 years.

Prior exposure to at least one ITP-directed therapy (e.g., corticosteroids, intravenous immunoglobulin, recombinant human thrombopoietin, TPO-RAs, immunosuppressants, or splenectomy), including a minimum 4-week course of an oral TPO-RA (hetrombopag or eltrombopag) that was discontinued due to insufficient response.

Platelet count < 30 × 10⁹/L at screening, OR platelet count < 50 × 10⁹/L with concurrent clinically significant bleeding.

Stable glucocorticoid dose (e.g., prednisone or methylprednisolone, not exceeding 4 tablets daily) for at least 2 weeks, and stable dosing of any other immunosuppressants for at least 4 weeks prior to enrollment.

No receipt of intravenous immunoglobulin within 2 weeks before the first dose of study treatment.

No platelet transfusion within 1 week before the first dose of study treatment.

Exclusion Criteria:

Secondary ITP due to underlying conditions such as other autoimmune disorders, viral infections, or drug exposure.

Presence of active malignancy, pregnancy, significant cardiovascular or cerebrovascular disease, or history of arterial/venous thrombosis.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy evaluation | from week 2 to month 12
  Efficacy assessments (platelet count) are performed weekly from Week 2 to Week 8, and then monthly until Month 12. Efficacy evaluation relies on time to platelet response, overall response rate, complete response rate and maintained response rate
Incidence of severe Adverse Events | up to 12 months
  Adverse events include the monitoring of the incidence of thrombotic events, myelofibrosis, and severe infections.

SECONDARY OUTCOMES:
Long-term Sustained Response Rate versus Relapse Rate | at 6 months and 12 months
Proportion of Participants Achieving a Rapid Platelet Response | within the first 8 weeks of treatment
  Platelet count is assessed weekly during this period
Change in Bleeding Score Over Time | up to 12 months
Incidence of other adverse events | up to 12 months
  Recording the incidence of other adverse events, such as liver and kidney dysfunction, and hypersensitivity reactions.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China